CLINICAL TRIAL: NCT01067508
Title: Effects of Naturally Occurring Silicon in Drinking Water on Bone Metabolism
Brief Title: Effects of Naturally Silicon-Rich Water on Bone Metabolism in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06-12-097-03
Record Dates: First submitted 2010-02-08; First posted 2010-02-11 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-05

CONDITIONS: Bone Diseases, Metabolic
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fiji Water (Experimental): Participants are asked to consume one liter of this silicon-rich water daily for three months.
  Interventions: Other: Fiji Water
- Aquafina Water (No Intervention): Participants are asked to drink one liter of this deionized water daily for three months.

INTERVENTIONS:
Other: Fiji Water — Participants are asked to drink one liter of this silicon-rich water daily for three months.
  Arms: Fiji Water

SUMMARY:
The aim of this research study is to determine by laboratory analyses the effects of drinking silicon-rich water on bone health. This will be determined from blood and urine samples from subjects who will be asked to drink 1 liter per day of either silicon-rich water or water without silicon for 12 weeks.

DETAILED DESCRIPTION:
Naturally occurring silicon as aqueous silicic acids at a level of 85 mg/liter which is well within safe intake limits occurs in water obtained from artesian wells in Fiji (Fiji Water, Inc.). Other drinking waters (e.g. Aquafina, Crystal Geyser, etc.) have all trace minerals including silicon removed by reverse osmosis. Silicon may be a necessary mineral for bone health. Therefore, this study aims to demonstrate the potential beneficial effects of short-term intake of silicon-rich water (85 mg/day of silicon in the diet from 1 liter of Fiji Water) compared to deionized water (with no silicon) over 12 weeks in normal postmenopausal women. The women to be studied will be stratified by bone density (based on T score by DEXA) and have analyses of biomarkers of bone metabolism to achieve the following specific aims:

1. To conduct a prospective randomized controlled trial in two mixed groups of 15 normal postmenopausal women and osteopenic pre- and peri-menopausal women receiving either 1 liter per day of FIJI water (A) or 1 liter per day of purified drinking water with no minerals (B). During screening we will ask prospective participants about their menopausal status (where post-menopausal means having no menstrual period for one year), block on their menopausal status, and randomize to either Treatment A or Treatment B. There will be 7-8 post-menopausal women and 7-8 pre- or peri-menopausal women in each group.
2. To determine silicon absorption by measuring urinary silicon excretion
3. To determine bone resorption and turn over markers by measuring urinary N-Telopeptide, serum bone alkaline phosphatase, osteocalcin, procollagen Type I Intact N-Terminal Propeptide, 25 hydroxyvitamin D, parathyroid hormone (PTH) and calcium.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) < 30
* Postmenopausal women with no evidence of osteoporosis by dual energy X-ray absorptiometry (DEXA) scan (T ≥ -2 in the total hip and lumbar spine).
* Pre- or peri-menopausal women with osteopenia but no evidence of osteoporosis by DEXA scan (-1.5 ≤ T ≤ -2 in the total hip and lumbar spine)
* No estrogens or corticosteroids
* No prior history of bisphosphonate medication
* Otherwise in good health with no significant illnesses which could affect bone metabolism such as hypercortisolism, untreated hypothyroidism, treatment with statins or other drugs affecting bone metabolism other than calcium and vitamin D3.
* No change in exercise regimen or calcium intake in the past 3 months.
* Subject must sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or randomization. A subject will be excluded for any condition that might compromise the ability to give truly informed consent for participation in the study.

Exclusion Criteria:

* Males
* Premenopausal women with DEXA T scores ≥ -1.5 or ≤ -2.
* Postmenopausal women with DEXA T scores ≤ -2.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Heber, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Z, Karp H, Zerlin A, Lee TY, Carpenter C, Heber D. Absorption of silicon from artesian aquifer water and its impact on bone health in postmenopausal women: a 12 week pilot study. Nutr J. 2010 Oct 14;9:44. doi: 10.1186/1475-2891-9-44. PMID 20946656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited by posting flyers around the UCLA campus community. Initial eligibility will be determined by a telephone conversation in which the study procedures and inclusion/exclusion criteria are reviewed.
Groups:
- Fiji Water: Participants are asked to consume 1 liter of this silicon-rich water daily for 12 weeks.
- Aquafina Water: Participants are asked to drink 1 liter of this deionized water daily for 12 weeks.
Period: Overall Study
Arm/Group | Fiji Water | Aquafina Water
Started | 10 | 9
Completed | 10 | 7
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Fiji Water: Participants are asked to consume 1 liter of this silicon-rich water (Fiji) daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Fiji Water | Aquafina Water | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (6.5) | 54.4 (3.9) | 53.75 (5.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Silicon Absorption at 12 Weeks
Description: Change from baseline in silicon absorption in response to silicon-rich water (Fiji) supplementation for 12 weeks was determined by measuring urinary solicon concentration (mg/mg) normalized to creatinine.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: mg/mg creatinine
Groups:
- Fiji Water: Participants are asked to drink 1 liter of this silicon-rich water daily for 12 weeks.
Arm/Group | Aquafina Water | Fiji Water
Number analyzed (Participants) | 9 | 10
mg/mg creatinine
  baseline silicon | 0.010 (0.004) | 0.016 (0.01)
  12 week silicon | 0.009 (0.006) | 0.037 (0.014)
Statistical Analysis 1: Comparison: Fiji Water; Comparison was made to 12 weeks minus baseline change in Fiji water group; Test type: Other; p = 0.003, t-test, 2 sided — p<0.05 was defined as significant
Statistical Analysis 2: Comparison: Aquafina Water; Comparison was made to the 12 week minus baseline change in Aquafina (control) group; Test type: Other; p = 0.68, t-test, 2 sided — p<0.05 was defined as significant

ADVERSE EVENTS:
Groups:
- Fiji Water: Participants are asked to consume 1 liter of this silicon-rich water (Fiji) daily for three months.
Arm/Group | Fiji Water | Aquafina Water
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fiji Water (N=10) | Aquafina Water (N=9)
Cardiovascular Health (Cardiac disorders) | 0 (0) | 1 (1) — One subject was withdrawn by the investigator concerning her cardiovascular health (not specified).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes